CLINICAL TRIAL: NCT06789042
Title: Efficacy of Perineural Dexamethasone to Prolong Anesthesia After Erector Spinae Plane Block for Total Hip Arthroplasty
Brief Title: Dexamethasone for ESPB in Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/2024
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Arthritis
Keywords: erector spinae plane block; total hip arthroplasty; pain management; perineural adjuvant
MeSH Terms: conditions — Osteoarthritis, Hip; Agnosia | interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Ultrasound-guided ESPB - 20ml 0,2% ropivacaine + 2ml 0.9% NaCl
  Interventions: Drug: 0.9%NaCl
- Dexamethasone (Active Comparator): Ultrasound-guided ESPB - 20ml 0,2% ropivacaine + 4mg Dexamethasone
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: 0.9%NaCl — 20ml 0.2% Ropivacaine + 2.0ml 0.9% NaCl
  Arms: Control group
Drug: Dexamethasone 4mg — 20ml 0.2% Ropivacaine + 4mg Dexamethasone
  Arms: Dexamethasone

SUMMARY:
Effect of adding Dexamethasone to Erector Spinae Plane Block in Patients undergoing Total Hip Arthroplasty

DETAILED DESCRIPTION:
Hip arthroplasty is one of the most common orthopaedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prostheses. Regional anaesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total hip arthroplasty
* patients aged >65 and <100 years
* patients able to provide informed consent
* patients able to reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a language barrier

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Total Opioid Consumption | 48 hours after procedure
  otal opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Nerve damage [range 0-4] | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
blood glucose | 12 hours after surgery
  blood glucose levels
blood glucose | 24 hours after surgery
  blood glucose levels
blood glucose | 48 hours after surgery
  blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Resyner, MD PhD, Study Director — Poznań University of Medical Science
Locations (1):
- Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No